CLINICAL TRIAL: NCT07041554
Title: Examination of Cardiovascular Risk Factors and Physical Activity in Chronic Kidney Patients Treated With Peritoneal Dialysis
Brief Title: Cardiovascular Risk Factors and Physical Activity in Chronic Kidney Patients on Peritoneal Dialysis
Status: Not yet recruiting | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ayten Demir, Graduate Student, Dokuz Eylul University
Other Study IDs: DEU-FTR-AE-02
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases; Cardiovascular Risk Factors; Arterial Stiffness; Physical Activity
Keywords: cardiovascular risk factors; physical activity; arterial stiffness; accelerometer; peritoneal dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Kidney Disease Patients Treated with Peritoneal Dialysis: The study will examine cardiovascular risk factors and physical activity parameters in a sample of 23 participants.

SUMMARY:
The objective of this study was to examine the association between cardiovascular risk factors and physical activity parameters in patients with chronic kidney disease who are treated with peritoneal dialysis.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is defined as a progressive disease in which kidney function is permanently impaired for a period of at least three months, glomerular filtration rate falls below 60 milliliters per minute per 1.73 square meters of body surface area, and the kidneys are structurally or functionally damaged. As the kidneys' capacity to regulate fluid, electrolyte, and acid-base balance decreases substantially in the later stages of CKD, renal replacement therapy is necessary to maintain renal function. Peritoneal dialysis, a type of renal replacement therapy, involves the use of a specialized dialysis solution that is injected into the abdominal cavity to effectively remove waste materials and excess fluids from the body.

The risk of cardiovascular disease is higher in peritoneal dialysis (PD) patients compared to the general population. Therefore, it is critical to identify these risk factors and develop effective interventions to reduce the risk of mortality, increase adherence to treatment, and improve quality of life. Arterial stiffness, a pivotal factor, has been shown to markedly elevate the risk of cardiovascular disease in PD patients and is associated with fluid overload and vascular calcification.

Physical activity plays a significant role in the reduction of cardiovascular risk factors in patients with PD. Regular exercise has been shown to improve cardiovascular health, control obesity, lower blood pressure, improve lipid profile, enhance insulin sensitivity, and increase overall physical activity levels. Consequently, these factors contribute to a reduction in cardiovascular disease (CVD) risk in PD patients. A notable study has concluded that physical activity plays a pivotal role in cardiovascular health and possesses the potential to reduce the risk of cardiovascular disease (CVD) in kidney transplant patients. Notably, studies have highlighted that physical activity levels in peritoneal dialysis patients are often suboptimal due to socio-demographic factors, fatigue, pain, psychological problems, and a lack of knowledge about exercise. This underscores the need for further research in this area to elucidate effective strategies for promoting physical activity and enhancing cardiovascular health in PD patients.

The present study will include individuals with chronic kidney disease who are followed up by the Nephrology Outpatient Clinic of Dokuz Eylül University Research and Application Hospital and treated with peritoneal dialysis. The objective of the study is to examine the relationship between cardiovascular risk factors and physical activity parameters in chronic kidney disease patients treated with peritoneal dialysis. Patients who meet the specified criteria will be included in the study. A comprehensive collection of sociodemographic and clinical information will be conducted, followed by an evaluation of cardiovascular risk factors. Heart rate, blood pressure, waist circumference, body mass index, laboratory findings (lipid profile [total cholesterol level, LDL and HDL cholesterol, triglycerides], fasting glucose value, HbA1C value, hemoglobin, CRP, proteinuria, glomerular filtration rate (GFR)), smoking history, and risk percentage will be determined with the HeartScore scoring system. The IEM Mobil-O-Graph® device will be used for arterial stiffness measurement. The physical activity parameters will be evaluated using an accelerometer (Sensewear Armband device), and the relationship between them will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic kidney disease
* Peritoneal dialysis treatment for at least three months
* Age ≥ 18

Exclusion Criteria:

* Mini Mental Test Score < 24
* Serious cardiovascular, pulmonary, or neurological conditions that make it impossible to wear an accelerometer
* Inability to walk independently
* Conditions affecting participation in daily life due to lower limb injury or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease who are followed up by the Nephrology Outpatient Clinic of Dokuz Eylül University Research and Application Hospital and treated with peritoneal dialysis will be included in the study.
Sampling Method: Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2025-06-23 (Estimated); Primary Completion 2025-09-02 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Physical Activity Level | Seven days
  Physical activity is defined as any body movement that results in the body expending more energy than its basal level of energy expenditure, due to skeletal muscle contraction. The assessment of physical activity levels will be conducted using the SenseWear Armband (SWK). The SWK will be used to obtain several pieces of information, including the number of steps, total energy expenditure (in calories), average day and night sleep time (in minutes), average day and night reaching time (in minutes), average metabolic equivalent (MET), active energy expenditure (in calories) consumed during moderate (3 MET) physical activity, and physical activity duration (in minutes, 3 MET). Subjects will be requested to utilize the device for a period of seven consecutive days.
Arterial Stiffness Measurement | 1 day
  Arterial stiffness represents the viscoelastic properties of the vessel wall, indicates vascular damage, and is a measure of the degree of atherosclerosis. Increased arterial stiffness or decreased compliance indicates diffuse atherosclerotic involvement of the vasculature. One of the non-invasive techniques used to assess arterial stiffness is pulse wave analysis (PWA). PWA examines the pressure waveforms in the major arteries. Pulse wave velocity (PWV) and amplification index (Alx) are indices of arterial stiffness.PWV is the velocity of the pulse propagating along the arterial segment. Alx is the ratio of the difference between the late systolic pressure reflected from the periphery and the early systolic pressure to the pulse pressure and is expressed as a percentage. The IEM Mobil-O-Graph® device is used to assess arterial stiffness.
Assessment of Cardiovascular Risk Factors | 1 day
  The following health metrics will be evaluated using the HeartScore scoring system to determine risk percentage: heart rate, blood pressure, waist circumference, body mass index, lipid profile (total cholesterol level, LDL and HDL cholesterol, triglycerides), fasting glucose value, HbA1C value, hemoglobin, CRP, proteinuria, smoking history, and glomerular filtration rate (GFR).The HeartScore system is a web-based risk prediction and management program that aims to support clinicians in optimizing individual cardiovascular risk reduction. The HeartScore web-based program utilizes a sophisticated algorithm to calculate the 10-year cardiovascular mortality risk based on age, gender, smoking habits, blood pressure, blood cholesterol, and the total cholesterol/HDL ratio. The European (High and Low) and National versions are currently available. However, the program is designed by national cardiology associations to be adapted to the local conditions of the countries.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Faculty of Physical Therapy and Rehabilitation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The reason for not sharing data is the concern about unauthorized use.